CLINICAL TRIAL: NCT02444819
Title: A Multicenter, Single-arm, Phase II Exploratory Trial to Evaluate the Efficacy and Safety of HM61713 as the 1st-line Anticancer Agent in NSCLC Patients With EGFR Mutation
Brief Title: Phase II Trial to Evaluate the Efficacy and Safety of HM61713 as the 1st-line NSCLC Anticancer Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-EMSI-201
Record Dates: First submitted 2015-05-12; First posted 2015-05-15 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: HM61713; Epidermal Growth Factor Receptor mutation positive NSCLC; olmutinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — olmutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HM61713 (Experimental): Subjects who entered the study will be administered HM61713 800 mg per day.
  Interventions: Drug: HM61713

INTERVENTIONS:
Drug: HM61713 — HM61713 will be administered to evaluate efficacy and safety of subjects.
  Other Names: Olmutinib

SUMMARY:
A multi-center, single-arm. Phase 2 exploratory trial to evaluate the efficacy and safety of HM61713 as the 1st-line anticancer agent in none-small cell lung cancer patients with EGFR mutation

DETAILED DESCRIPTION:
HM-EMSI-201 study targets NSCLC patients with EGFR mutations by HM61713 anticancer drug as the first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 19 years at the time of signing informed consent
* Cytologically or histologically confirmed, advanced or metastatic NSCLC which is not amenable to curative surgery (Stage IIIb or IV)
* Documented EGFR mutations (excluding exon 20 insertion)
* At least one lesion that can be used as a measurable lesion per RECIST version 1.1
* Performance status under 1 per ECOG score
* Life expectancy of at least 12 weeks
* Adequate hematological and biological functions
* Provide voluntary consent to participate the study and sign the written consent form

Exclusion Criteria:

* Treatment of chemotherapy, biological therapy or immunotherapy for anticancer therapies of stage IIIb or IV NSCLC (excluding adjuvant/neoadjuvant chemotherapy, radiotherapy or radiochemotherapy prior to more than 6 months from the first dose of study treatment
* History of treatment with an EGFR targeting small molecule or antibodies
* Any non-study related significant surgical procedures requires general anesthesia or breathing apparatus within the past 4 weeks of the first dose of study treatment (excluding video-assisted thoracoscopic surgery or open-and-closed surgery prior to the past 2 weeks of the first dose of study treatment)
* History of any other malignancy within 5 years of study participation (other than curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors unless it has been definitively treated with no evidence of relapse or recurrence within the past 3 years)
* Clinically significant uncontrolled conditions of infectious disease including active infection that requires parenteral antibiotics (except when conditions are definitively treated or controlled)
* Spinal cord compression, leptomeningeal carcinomatosis, symptomatic or uncontrolled brain metastasis
* Presence or history of ILD or pulmonary fibrosis
* NYHA class III or IV cardiac insufficiency, uncontrolled hypertension, experienced unstable angina pectoris or cardiac infarction within 6 months, uncontrolled cardiac arrhythmia or clinically significant abnormal cardiovascular activities
* LVEF < 40%
* Presence or history of pancreatitis or serum amylase > 1.5xULN
* Inability to swallow the formulated product or gastrointestinal tract abnormalities which would preclude administration or absorption of study medication
* Mental or congenital disabilities (e.g. dementia or epilepsy) which would preclude understanding of informed consent or following the study protocol
* History of hypersensitivities to investigational drug or related similar class drugs
* Pregnant or breast feeding
* Unwillingness of adequate contraception during study treatment and at least 2 months after treatment
* Unwillingness of following procedures of study protocol or follow-up assessments; Unable to follow up for long term for psychological, social, family problem or geographical reasons
* History of treatment with other investigational drugs or investigational medical devices prior to 28 days of the first dose of study treatment
* In the opinion of the investigator, the patient is an unsuitable candidate to the study
* ECG finding of QTcF > 450 msec at rest

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-03; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate | At baseline and every 6 weeks until disease progression or withdrawal from study, expected average 1 year
  To obtain a assessment of anti-tumor activity of HM61713 by evaluation of tumor response using RECIST version 1.1

SECONDARY OUTCOMES:
Progression-free survival | At baseline and every 6 weeks until disease progression or withdrawal from study, expected average 1 year
  To obtain a assessment of anti-tumor activity of HM61713 by evaluation of tumor response using RECIST version 1.1
Disease control rate | At baseline and every 6 weeks until disease progression or withdrawal from study, expected average 1 year
  To obtain a assessment of anti-tumor activity of HM61713 by evaluation of tumor response using RECIST version 1.1
overall survival | At baseline and every 6 weeks until disease progression or withdrawal from study, expected average 1 year
  To obtain a assessment of anti-tumor activity of HM61713 by evaluation of tumor response using RECIST version 1.1
Time to progression | At baseline and every 6 weeks until disease progression or withdrawal from study, expected average 1 year
  To obtain a assessment of anti-tumor activity of HM61713 by evaluation of tumor response using RECIST version 1.1
Maximum decrease in tumor size | At baseline and every 6 weeks until disease progression or withdrawal from study, expected average 1 year
  To obtain a assessment of anti-tumor activity of HM61713 by evaluation of tumor response using RECIST version 1.1
Quality of life questionnaire | At baseline and every visit, expected average 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yohan Kim, MD, Study Director — Hanmi Pharmaceutical Company Limited; Keunchil Park, MD PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Seoul, South Korea